CLINICAL TRIAL: NCT07321119
Title: Correlation Between Endurance and Proprioception Function in Cervical Radiculopathy
Brief Title: Correlation Between Cervical Deep Flexors Endurance and Proprioception Function in Cervical Radiculopathy
Status: Not yet recruiting | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Ibrahim Ahmed Ibrahim Abu Ella, Lecturer, Delta University for Science and Technology
Other Study IDs: trial registry 3
Record Dates: First submitted 2025-12-13; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: cevical range of motion device — Cervical proprioception was evaluated using the Cervical Range of Motion (CROM) device by assessing joint position sense (JPS). With the participant seated in an upright position, the CROM device was securely fitted to the head. The patient was instructed to actively move the head from a neutral starting position into a specific direction (flexion, extension, rotation, or lateral flexion), then return to the perceived neutral position with eyes closed.
  The difference between the starting neutral position and the repositioned angle was recorded as the joint position error (JPE), measured in degrees. Multiple trials were performed for each movement direction, and the mean JPE value was calculated. Higher JPE values indicated poorer cervical proprioceptive accuracy. The CROM device is considered a reliable and valid clinical tool for quantifying cervical proprioception in patients with cervical radiculopathy.

SUMMARY:
In cervical radiculopathy, reduced endurance of the deep cervical flexor muscles is associated with impaired cervical proprioception. This relationship reflects altered sensorimotor control due to muscle dysfunction and neural compromise, emphasizing the need for deep flexor endurance training in rehabilitation.

DETAILED DESCRIPTION:
In patients with cervical radiculopathy, endurance of the deep cervical flexor muscles (longus capitis and longus colli) plays a crucial role in maintaining cervical segmental stability and accurate sensorimotor control. These muscles are rich in muscle spindles and provide continuous afferent input necessary for cervical proprioception, including joint position sense and movement accuracy. When deep cervical flexor endurance is reduced, there is increased reliance on superficial neck muscles, leading to altered motor patterns and diminished quality of proprioceptive feedback.

Cervical radiculopathy further disrupts proprioceptive function through nerve root compression, inflammation, and impaired neural conduction, which affect both sensory input and motor output. This neuromuscular dysfunction results in increased joint position errors, delayed muscle activation, and poor postural control. Consequently, a significant correlation is observed between decreased deep cervical flexor endurance and impaired cervical proprioception, suggesting that deficits in muscle endurance contribute directly to sensorimotor dysfunction. These findings support rehabilitation approaches that emphasize endurance training of the deep cervical flexors to restore proprioceptive accuracy and cervical motor control in patients with cervical radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with cervical radiculopathy based on clinical examination (± imaging confirmation).

Presence of neck pain with radiating symptoms to the upper limb for at least 4 weeks.

Age range 20-60 years.

Ability to understand instructions and participate in cervical endurance and proprioception assessments.

Exclusion Criteria:

* History of cervical spine surgery or acute cervical trauma.

Presence of neurological disorders other than cervical radiculopathy (e.g., stroke, multiple sclerosis).

Vestibular disorders or conditions affecting balance and head position sense.

Inflammatory, rheumatologic, or severe musculoskeletal conditions involving the cervical spine.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consisted of 80 patients with cervical radiculopathy recruited from outpatient physical therapy clinics. Participants were adults of both sexes, aged between 20 and 60 years, presenting with neck pain associated with unilateral or bilateral upper limb radicular symptoms, including pain, numbness, or weakness. Cervical radiculopathy was diagnosed based on clinical examination findings such as dermatomal pain distribution, positive cervical compression tests, and neurological deficits, with imaging confirmation when available.
  All participants were in the subacute to chronic stage of the condition and were able to sit independently and follow verbal instructions during assessment. Patients with a history of cervical spine surgery, recent trauma, vestibular disorders, or other neurological or systemic conditions affecting cervical proprioception were excluded. This population was selected to investigate the relationship between cervical deep flexor endurance and cerv
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Cervical proprioception errors by using joint position sense via CROM device | baseline
  Cervical proprioception was assessed using the CROM device by measuring joint position sense error. Participants were seated upright with the trunk stabilized and the CROM mounted on the head; visual input was eliminated by closing the eyes. From a neutral head position, participants actively moved the head to a predetermined target angle (approximately 50-60% of available cervical range of motion) in flexion, extension, or rotation, held the position briefly, returned to neutral, and then attempted to reproduce the target position. The absolute difference between the target and reproduced angles, recorded in degrees by the CROM, represented the joint position error, and the mean of three trials for each movement direction was used for analy

SECONDARY OUTCOMES:
Deep flexor cervical muscle endurance using biofeedback device | baseline
  Deep cervical flexor muscle endurance was assessed using a pressure biofeedback unit. Participants were positioned in crook-lying with the pressure cuff placed suboccipitally and inflated to a baseline pressure of 20 mmHg. After instruction and practice of the craniocervical flexion action, participants were asked to incrementally increase and maintain pressure (22-30 mmHg) by performing a gentle nodding movement without activation of superficial neck muscles. Endurance was recorded as the maximum pressure level that could be held steadily for 10 seconds with correct technique, and the total performance score was determined based on the highest successfully maintained pressure level.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rafiq S, Zafar H, Gillani SA, Waqas MS, Liaqat S, Zia A, Rafiq Y. Effects of Neurodynamic Mobilization on Health-Related Quality of Life and Cervical Deep Flexors Endurance in Patients of Cervical Radiculopathy: A Randomized Trial. Biomed Res Int. 2022 Oct 5;2022:9385459. doi: 10.1155/2022/9385459. eCollection 2022. PMID 36246968